CLINICAL TRIAL: NCT03287154
Title: Interest of tDCS in Help for Supporting Alcohol Abstinence
Acronym: ITAMAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-A00304-47
Record Dates: First submitted 2017-09-07; First posted 2017-09-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Alcoholic Intoxication
Keywords: Alcohol Abstinence; Alcohol Addiction; Alcohol Consumption; Alcohol Dependence
MeSH Terms: conditions — Alcoholic Intoxication; Alcohol Abstinence; Alcoholism; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS stimulations (Experimental): Patients in this arm will receive 10 tDCS active stimulations of 2 mA (1 stimulation per day from Monday to Friday during 2 weeks).
  Interventions: Device: Active tDCS stimulations
- Sham tDCS (Sham Comparator): Patients in this arm will receive 10 sham stimulations (1 stimulation per day from Monday to Friday during 2 weeks).
  As soon as the power will have reached the maximal intensity as in the active arm, the stimulation will be stopped.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS stimulations — 20 min, 2mA
  Arms: Active tDCS stimulations
Device: Sham tDCS — 20 min, Sham
  Arms: Sham tDCS

SUMMARY:
The aim of the study is to evaluate in patients with alcohol disorder and forehand weaned the efficiency of 10 active tDCS sessions versus 10 sham (placebo) sessions in the support of abstinence at 3 months.

DETAILED DESCRIPTION:
The study takes place at one site (Henri Laborit Hospital, Poitiers, France) and is comparative, randomized and controlled.

There are 2 groups : one group is receiving sessions of active tDCS (active group) whereas the second group is receiving sham (placebo) sessions (control group).

Patients are randomized either in the active group or in the control group with a 1:1 ratio.

An unblinded investigator is responsible of the stimulation part and could not evaluate the patients. The other investigators are blinded and could evaluate the patients.

The study is going to evaluate the effect produces by stimulations in the two groups.

In the placebo group, after the intensity has reached its maximal intensity (the same as in the active group), the stimulation is stopped after few seconds (30 seconds in mostly studies). This process allow patients in the placebo group to feel the same sensations as patients in the active group (indeed, tingles and itches are felt only during the first few seconds of stimulation). The poor duration of stimulation do not produces clinical effect.

The study begins after a withdrawal period of 7 days +/- 3 days with 10 stimulations of 2 mA during 20 minutes from Monday to Friday during 2 weeks.

Following these stimulation sessions, the patient will have 5 follow-up visits on site with an investigator and 2 phone follow-up.

Visits:

* Pre-inclusion visit
* V0 visit (inclusion visit): takes place at the earliest 48 hours after stopping benzodiazepines used in the withdrawal period.
* Treatment (weeks 0 and 1): 5 days of treatment per week during 2 weeks 2 arms : sham (placebo, 10 stimulations) vs active (10 stimulations of 2 mA)
* Visit 1 (Week 4) : short nurse consultation
* Visit 2 (Week 6) : short medical consultation
* Visit 3 (Week 10) : short medical consultation
* Visit 4 (Week 14) : long medical consultation
* Visit 5 (Week 18) : nurse phone follow-up
* Visit 6 (Week 22) : nurse phone follow-up
* Visit 7 (Week 26) : long medical consultation

ELIGIBILITY:
Inclusion Criteria:

* patient aged from 18 to 70 years old
* patient free, without guardianship
* absence of epileptic pathology
* patient affiliated to the french health security or benefiting through a third party
* signed informed consent after having received a clear and honest information on the study.
* patient with a disorder linked to the use of alcohol (define by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) classification) clinically evaluated.
* patient requesting for an alcohol withdrawal
* patient able to read and write

Exclusion Criteria:

* patient not affiliated to the french health security or not benefiting through a third party
* woman in reproductive capacity without effective contraception (hormonal/mechanical: per os, injectable, transcutaneous, implantable, intra-uterine device or chirurgical: tubal ligation, hysterectomy, total ovariectomy) or breastfeeding
* patient hospitalized under duress
* patient with guardianship
* somatic complications during the alcohol withdrawal phase
* current psychiatric decompensation (mood disorder, suicide risk, psychotic disorders).
* patient under benzodiazepines treatment
* patient with scalp cutaneous lesion
* history of cranial traumatism
* patient with intra-cerebral metallic object
* patient with a pacemaker
* epileptic pathology
* patient in emergency condition or unable to give personally her/his consent
* another dependence other than alcohol or tobacco
* mental illness syndrome and Korsakoff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Alcohol Abstinence | 3 months
  The primary outcome is to evaluate the interest of the transcranial Direct Current Stimulation (tDCS) for helping the abstinence support in addictive alcoholic patients.

SECONDARY OUTCOMES:
Relapse control | 6 months
  Evaluation of tDCS interest in help for relapse control.
Alcohol consumption | 6 months
  Impact on alcohol consumption based on the Total Alcohol Consumption (TAC).
Anxiety-depression | 6 months
  Impact on the anxiety-depression symptomatology
Tobacco consumption | 6 months
  Impact on tobacco consumption (decrease of cigarette consumption).
Safety assessment with adverse and/or intercurrent events analysis. | 6 months
  The clinical tolerability will be objectified through the analysis of adverse and /or intercurrent events occuring all along the study. Theses events will be assessed at every study visit during patient examination.
Cognitive functions assessments with the Moca-test questionnaire. | 6 months
  The score to the Moca-test will permit to assessed the cognitive functions from baseline (week 0) to the week 14 and from baseline from the week 26.
Executive functions assessments with the scale Barratt Impulsiveness Scale (BIS 11). | 6 months
  This examination will be assessed from week 0 to Day 9, from week 0 to week 14 and from week 0 to week 26.
Executive functions assessments with the Go NoGo task. | 6 months
  This examination will be assessed from week 0 to Day 9, from week 0 to week 14 and from week 0 to week 26.
Executive functions assessments with the Wisconsin Card Sorting Test (WCST). | 6 months
  This examination will be assessed from week 0 to Day 9, from week 0 to week 14 and from week 0 to week 26.
Executive functions assessments with the Stroop test. | 6 months
  This examination will be assessed from week 0 to Day 9, from week 0 to week 14 and from week 0 to week 26.
Executive functions assessments with the IOWA Gambling Task (IGT). | 6 months
  This examination will be assessed from week 0 to Day 9, from week 0 to week 14 and from week 0 to week 26.

CONTACTS AND LOCATIONS:
Overall Officials: Nematollah Jaafari, Professor, Principal Investigator — Centre Hospitalier Henri Laborit
Locations (2):
- France (2):
  - Centre Hospitalier Henri Laborit, Poitiers
  - Centre Hospitalier Nord-Deux-Sèvres, Thouars

IPD SHARING:
Plan to Share IPD: No